CLINICAL TRIAL: NCT00475878
Title: Antidepressants During Office-Based Buprenorphine
Brief Title: SSRI and Buprenorphine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Michael Stein, MD, Principal Investigator, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA022207; 0807-002
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Results first posted 2012-04-03 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Opiate Dependence; Depression
Keywords: opiate use; depression; buprenorphine; escitalopram
MeSH Terms: conditions — Opioid-Related Disorders; Depression | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- escitalopram (Active Comparator)
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — 10mg escitalopram/day for 3 months
  Arms: escitalopram
Drug: placebo — placebo capsule/day for 3 months
  Arms: placebo

SUMMARY:
This study is designed to test whether treatment of depressive symptoms using escitalopram improves adherence to Buprenorphine and reduces symptoms of depression for individuals receiving Buprenorphine through their medical provider.

DETAILED DESCRIPTION:
Participants interested in receiving Buprenorphine will be offered the opportunity to enroll in this study. Enrolled study participants will complete interviews at baseline and again every two weeks for a total of 8 interviews over 3 months. In this double-blind randomized controlled trial, participants will either receive a placebo or escitalopram (10mg). All participants will also be followed by their Buprenorphine clinic medical provider. Questions during the face-to-face interviews will assess mood, drug craving, pain, sleep, medication adherence and drug-related experiences. Comparison(s): Participants randomized into the medication component of the study as compared to participants randomized into the placebo component of the study.

ELIGIBILITY:
Inclusion Criteria:

* opiate dependence
* Ham-D > 14

Exclusion Criteria:

* no psychiatric contraindications to using escitalopram
* no medical contraindications to using escitalopram
* methadone dose < 30
* no current SSRI use

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2006-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Stein, M.D., Principal Investigator — Rhode Island Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Tsui JI, Anderson BJ, Strong DR, Stein MD. Craving predicts opioid use in opioid-dependent patients initiating buprenorphine treatment: a longitudinal study. Am J Drug Alcohol Abuse. 2014 Mar;40(2):163-9. doi: 10.3109/00952990.2013.848875. Epub 2014 Feb 12. PMID 24521036
- [Derived] Cioe PA, Anderson BJ, Stein MD. Change in symptoms of erectile dysfunction in depressed men initiating buprenorphine therapy. J Subst Abuse Treat. 2013 Nov-Dec;45(5):451-6. doi: 10.1016/j.jsat.2013.06.004. Epub 2013 Jul 23. PMID 23891461
- [Derived] Strong DR, Brown RA, Sims M, Herman DS, Anderson BJ, Stein MD. Persistence on a stress-challenge task before initiating buprenorphine treatment was associated with successful transition from opioid use to early abstinence. J Addict Med. 2012 Sep;6(3):219-25. doi: 10.1097/ADM.0b013e31825d927f. PMID 22864399
- [Derived] Tsui JI, Herman DS, Kettavong M, Anderson BJ, Stein MD. Escitalopram is associated with reductions in pain severity and pain interference in opioid dependent patients with depressive symptoms. Pain. 2011 Nov;152(11):2640-2644. doi: 10.1016/j.pain.2011.08.011. Epub 2011 Sep 15. PMID 21924552
- [Derived] Tsui JI, Herman DS, Kettavong M, Anderson BJ, Stein MD. Chronic pain and hepatitis C virus infection in opioid dependent injection drug users. J Addict Dis. 2011 Apr;30(2):91-7. doi: 10.1080/10550887.2011.554775. PMID 21491290
- [Derived] Stein MD, Herman DS, Kettavong M, Cioe PA, Friedmann PD, Tellioglu T, Anderson BJ. Antidepressant treatment does not improve buprenorphine retention among opioid-dependent persons. J Subst Abuse Treat. 2010 Sep;39(2):157-66. doi: 10.1016/j.jsat.2010.05.014. Epub 2010 Jul 3. PMID 20598836

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: placebo pill, daily for 12 weeks, for individuals entering buprenorphine treatment for opioid dependence
- 10 mg Escitalopram: 10 mg escitalopram pill, daily for 12 weeks, for individuals entering buprenorphine treatment for opioid dependence
Period: Overall Study
Arm/Group | Placebo | 10 mg Escitalopram
Started | 75 | 72
Completed | 75 | 72
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg Escitalopram | Total
Number analyzed (Participants) | 75 | 72 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 72 | 147
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.8 (9.8) | 38.3 (9.6) | 37.5 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 57 | 55 | 112
Region of Enrollment [Number; unit: participants]
  United States | 75 | 72 | 147

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Dropped Out of Buprenorphine Treatment
Description: Drop-out is defined as 7 or more days of missed Buprenorphine doses
Time Frame: 3 months
Population: Participants who were fully eligible for the study, completed the enrollment process and began study medication were used in an intent to treat analysis.
Measure: Number; unit: percentage of participants
Groups:
- 10 mg Escitalopram: in a double-blind, randomized controlled trial, participants were given 10mg escitalopram prior to buprenorphine induction
- Placebo: in a double-blind, randomized controlled trial, participants were given placebo prior to buprenorphine induction
Arm/Group | 10 mg Escitalopram | Placebo
Number analyzed (Participants) | 72 | 75
percentage of participants | 33.3 | 44.0
Statistical Analysis 1: Comparison: 10 mg Escitalopram vs Placebo; Test type: Superiority or Other; p = .19, Chi-squared; Odds Ratio (OR) = .64, 95% CI 2-sided [.33 to 1.24], Standard Error of Mean .22

2. Secondary Outcome: Depressive Symptoms
Description: Depressive symptoms, as measured by self-report during study interviews, using the Beck Depression Inventory II. Scores ranged from 0-63; higher scores indicate more depressive symptoms.
Time Frame: 3 months
Population: participants who were fully eligible for the study, completed the enrollment process and began study medication were included in an intent to treat analysis
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- 10 mg Escitalopram: individuals were given 10mg escitalopram prior to buprenorphine induction
- Placebo: individuals were given a placebo study medication prior to buprenorphine induction
Arm/Group | 10 mg Escitalopram | Placebo
Number analyzed (Participants) | 72 | 75
units on a scale | 12.31 (1.79) | 11.35 (1.46)
Statistical Analysis 1: Comparison: 10 mg Escitalopram vs Placebo; Test type: Superiority or Other; p = .18, t-test, 2 sided; Mean Difference (Final Values) = .96, 95% CI 2-sided [-2.79 to 5.84], Standard Error of Mean 2.16

ADVERSE EVENTS:
Time Frame: adverse event information was collected at each study appointment, which occurred every 1-2 weeks throughout participant's 12-week study participation.
Description: adverse event information was collected via structured questionnaires and by the study physician during bi-weekly medication visits.
Arm/Group | Placebo | 10 mg Escitalopram
Serious Adverse Events (participants affected / at risk) | 1/75 | 0/72
Other Adverse Events (participants affected / at risk) | 0/75 | 0/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=75) | 10 mg Escitalopram (N=72)
increasing clinical symptoms (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No